CLINICAL TRIAL: NCT06758206
Title: Effect of 10 Months of Flywheel Resistance Training Versus Traditional Resistance Training on Depressive Symptoms, Physical and Executive Function in Older Women With Sedentary Behaviors
Brief Title: Flywheel Resistance Training and Traditional Resistance Training in Older Women With Sedentary Behaviors
Acronym: FET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Vicosa (Other)
Responsible Party: Principal Investigator, Pablo Augusto Garcia Agostinho, Ph.D. Student in Physical Education, Principal Investigator, Federal University of Vicosa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.821.139
Record Dates: First submitted 2024-12-22; First posted 2025-01-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Depressive Symptoms; Physical Function; Executive Function; Resistance Training
Keywords: depressive symptoms; Physical Function; Executive function; Resistance training; Eccentric action; Older women
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Hidden and opaque envelope technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flywheel resistance training (Experimental): Flywheel resistance training will use the isoinertial multi-leg machine for lower and upper limbs for women.
  Interventions: Behavioral: Flywheel Resistance Training
- Traditional resistance training (Active Comparator): Traditional resistance training will use machines for the lower limbs and free weights for the upper limbs.
  Interventions: Behavioral: Traditional resistance training

INTERVENTIONS:
Behavioral: Flywheel Resistance Training — For each training session, 6 to 7 generic exercises will be performed, involving small and large muscle groups (leg extension, leg flexion, biceps curl, triceps extension, seated row, shoulder flexion and shoulder raise). They will perform 4 sets of 8 repetitions, with a 2-minute break between exercises and sets. They will perform these exercises at a high intensity (always 10 on the OMNI-RES Scale).
  Arms: Flywheel resistance training
Behavioral: Traditional resistance training — For each training session, 6 to 7 generic exercises will be performed, involving small and large muscle groups (leg extension, leg flexion, biceps curl, triceps extension, seated row, shoulder flexion and shoulder raise). They will perform 4 sets of 8 to 12 repetitions, with a 2-minute break between exercises and sets. They will perform these exercises at moderate and high intensities (6 to 10 on the OMNI-RES scale).
  Arms: Traditional resistance training

SUMMARY:
There are easily accessible and safe strategies, such as resistance training, that can contribute to reducing depressive symptoms and preserving physical and executive function in older women. Resistance training is defined as exercises performed either in water or on land, involving the use of a constant load or uniform weight, regardless of the training program. Various types of resistance training equipment are available, including free weights, pneumatic resistance machines, elastic bands, or even body weight. Specifically, eccentric muscle action occurs when the force applied to the muscle exceeds the momentary force produced by the muscle itself, resulting in the forced elongation of the muscle-tendon system during contraction.

To date, evidence from randomized clinical trials has compared the effectiveness of aerobic, resistance, and Pilates exercises in reducing depressive symptoms and improving physical and executive function in older women.

While experimental studies have demonstrated the efficacy of physical exercise, the effect of long-term eccentrically reinforced resistance training on depressive symptoms, physical function, and executive function in sedentary older women remains unclear.

Therefore, this study aims to evaluate the safety and effect of eccentrically reinforced resistance exercise versus traditional resistance training on depressive symptoms, physical and executive function, quality of life, different manifestations of muscle strength, body composition, vital signs, abdominal circumference, fall risk, and fatigue symptoms in sedentary older women over a 10-month period.

DETAILED DESCRIPTION:
Seventy Four older women will be randomly assigned to two groups: Flywheel resistance training and traditional resistance training. The interventions will be conducted at the Physical Education Department of the Federal University of Viçosa, with all sessions supervised by Physical Education professionals. Follow-up will be carried out through WhatsApp messages and phone calls. Both groups will train twice a week for 10 months. Participants in the experimental group will perform Flywheel resistance training on a multi-leg isoinertial machine targeting upper and lower body muscles, while the control group will use traditional machines and free weights. Each session will include 6 to 7 exercises, performed in 4 sets of 8 to 12 repetitions, with a 2-minute rest between sets and exercises. Training progression will be adjusted based on the participant's ability to exceed the maximum suggested repetitions with the same mobilized weight. Exercises will target various muscle groups, including leg extension, leg curl, bicep curl, tricep extension, seated row, shoulder flexion, and shoulder elevation.

Participants will be assessed at three time points during the training program: pre-intervention, 5 months, and 10 months after the intervention starts. Lower limb muscle strength will be evaluated using one-repetition maximum (1RM) tests on a knee extension machine and through maximal voluntary isometric contraction (MVIC), assessed with a load cell. Depressive symptoms will be measured using the Geriatric Depression Scale (GDS), validated for use in Brazil. Physical function will be assessed through the Timed Up and Go (TUG) test and the Senior Fitness Test (SFT). Executive function will be evaluated using the Victoria Stroop test, Digit Span (forward and backward), and the Trail Making Test (parts A and B). Quality of life will be assessed using the Brazilian version of the WHOQOL-Bref, while body composition will be analyzed through dual-energy X-ray absorptiometry (DXA). Blood pressure (systolic, diastolic, and mean arterial pressure) will be measured using an aneroid sphygmomanometer, and resting heart rate will be manually recorded after 3 minutes in a seated position. Abdominal circumference will be measured with a metal tape at the midpoint between the lower costal margin and the iliac crest, at the end of a normal expiration. Fall risk will be assessed using the Falls Efficacy Scale-International (FES-I) and the Berg Balance Scale. Fatigue symptoms will be evaluated using the Fatigue Symptom Inventory (FSI).

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older.
* Self-reported proficiency in speaking, writing, and understanding Portuguese.
* Willingness and availability to participate in all trial procedures.
* Good vision in at least one eye.
* Absence of any medical contraindications for engaging in physical exercise.
* Engage in less than 150 minutes of physical activity per week.
* Not clinical diagnosis of major depressive disorder at the time of the interventions.

Exclusion Criteria:

* Have uncontrolled chronic or psychiatric illnesses.
* Surgical procedures scheduled during the intervention period.
* Diagnosis of joint diseases such as osteoarthritis and arthrosis.
* Participating in aerobic or resistance exercise programs twice a week for the past three months.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Changes in baseline depressive symptoms at ten months. | Baseline, 5 and 10 months
  Test: The depressive state will be evaluated with a short version of the validated geriatric depression scale (GDS) in Brazil. There are 15 questions that inquire about feelings and a frequency that the person presents before certain conditions of life. These questions require categorical answers (yes or no). Of the 15 items, 10 indicate the presence of depression when answered positively. While the rest (1, 5, 7, 11 and 13) when answered negatively. A higher score indicates depression.
Change in baseline test Time up and go at ten months. | Baseline, 5 and 10 months
  Test: The time up and go will assess sitting balance, balance in transfers from sitting to standing, stability in ambulation and changes of direction. The test consists of the individual getting up from the chair, without arm support, walking 3 meters with safe and comfortable steps, without running, turning 180°, returning and sitting in the chair. The time taken to perform this task will be timed. Volunteers who perform the task in a time of less than 10 seconds will be considered with satisfactory mobility, for those who perform the test between 11 and 20 seconds will be classified with good mobility and for those who reach values greater than 20 seconds will be classified with mobility problems.
Change in baseline 30-s chair stand at ten months | Baseline, 5 and 10 months
  There will be a 30-s chair stand for the Senior Fitness Test (SFT), which is a battery of functional tests designed to assess the physical capacity needed for independence in older adults. This test assesses the number of repetitions an individual can lift from a chair in 30 seconds and evaluates leg strength. The more repetitions, the better the functionality.
Change in baseline 30-s arm curl at ten months | Baseline, 5 and 10 months
  The 30-s arm curl of the Senior Fitness Test (SFT) will be performed, which is a battery of functional tests designed to assess the physical capacity required for independence in older adults. This test evaluates the number of repetitions of bicep curls in 30 seconds with a weight of two kilos. It assesses arm strength. The more repetitions, the better the functionality.
Change in baseline 6-min walk at ten months | Baseline, 5 and 10 months
  The 6-min walk test will be carried out, which measures the distance covered in 6 minutes and assesses cardiovascular capacity. It is part of the Senior Fitness Test. The greater the distance covered, the better the functionality.
Change in baseline chair sit-and-reach at ten months | Baseline, 5 and 10 months
  The chair sit-and-reach test will be carried out, which measures the distance between the toes and the tip of the foot on an outstretched leg. It is part of the Senior Fitness Test. The shorter the distance between the limbs, the better the functionality.
Change in baseline back scratch at ten months | Baseline, 5 and 10 months
  The back scratch test will be carried out, which measures the distance between the middle fingers when reaching behind the back with both hands. It is part of the Senior Fitness Test. The shorter the distance between the limbs, the better the functionality.
Change in baseline 8-foot up-and-go at ten months | Baseline, 5 and 10 months
  The 8-foot up-and-go test will be carried out, which measures the time it takes to get up from a chair, walk 8 feet (2.4 m), turn around and return to the chair. It is part of the Senior Fitness Test. The shorter the time taken to complete the course, the better the functionality.
Change in Inhibitory control at ten months | Baseline, 5 and 10 months
  Test: Victoria Stroop test. Inhibitory control will be evaluated using the Victoria Stroop Test, which uses three tasks with 24 items each. The participant is evaluated according to how quickly she performs the task and the number of errors. The effect of interference is determined by calculating the extra time required to name the colors (of the printout) compared to the time required to name colors in the first control task (colors of the cards). The task performed faster indicates better performance.
Change in Working memory at ten months | Baseline, 5 and 10 months
  Working memory will be evaluated by Digit Span Forward and Backward. For the calculation of the test, the sum of the longest sequence of digits repeated, without error, over two trials in direct order is used.
Change in Cognitive flexibility at ten months | Baseline, 5 and 10 months
  Test composed of two parts (Tracks A and Tracks B). The execution time for each of the tests is limited to four minutes or three errors The test score will be obtained through the time spent to finish each part. For speed adjustment, the difference between the completion times of part B and part A will be calculated, in which smaller differences in scores indicate better speed adjustments.

SECONDARY OUTCOMES:
Change in baseline quality of life time at ten months. | Baseline, 5 and 10 months
  Test: World Health Organization Quality of Life Assessment Bref. The Brazilian version of the World Health Organization Quality of Life Assessment Bref will be utilized in this study. The 26 items produce 4 domains related to Quality of Life; physical (health), psychological, social relationships and environmental and an overall Quality of life and health satisfaction facet. Each item is measured from 1 to 5 on a Likert scale, with varying scale response anchors, where higher values represent higher Quality of life. One example of item is "How much do you enjoy life?", rated on the following response options (1) not at all, (2) a little, (3) a moderate amount, (4) very much, and (5) an extreme amount.
Maximum isometric voluntary contraction | Baseline, 5 and 10 months
  To evaluate the Maximum isometric voluntary contraction (MIVC) of the lower extremities, a load cell or extensiometric cell (MK®, CSL / ZL-1 T, MK Controle, Brazil) with a sampling frequency of 1000 Hz will be used.
1RM test | Baseline, 5 and 10 months
  To perform the one repetition maximum test (1RM), the knee extension exercise will be used on a BH fitness® Nevada Pro-t extension machine. To perform the test, the volunteer will be asked to extend the knee to form an angle of approximately 180° (final position) and return to the initial position.
Muscle power | Baseline, 5 and 10 months
  The evaluation of lower limb muscle power will be performed using the same knee extension machine used in the exercise sessions, starting from the same initial position (90º of kneeling flexion) and reaching the same final position (180º of knee extension) as the test of 1RM.
Change In Baseline Total body mass at ten months | Baseline, 5 and 10 months
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Change In Baseline lean mass At Ten Months | Baseline, 5 and 10 months
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Change In Baseline bone mineral content At Ten Months | Baseline, 5 and 10 months
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Change In Baseline bone mineral density At Ten Months | Baseline, 5 and 10 months
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Change In Baseline bone loss index throughout life At Ten Months | Baseline, 5 and 10 months
  Dual-engy X-ray absorptiometry (DXA) full body exam (GE Healthcare Lunar Prodigy Advance DXA System, software version 13.31).
Blood pressure | Baseline, 5 and 10 months
  Minimus® III aneroid tensiometer will be used, which has a maximum error margin of +/-3 mmHg. Systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean blood pressure (MBP) will be calculated. MBP will be obtained with the following mathematical operation: PAD + PAD + PAS / 3
Resting heart rate | Baseline, 5 and 10 months
  For Resting heart rate (HRR) measurement, women will be advised to sit for 3 minutes. After that moment, this variable will be taken manually in the radial or carotid pulse of the right side for 60 seconds.
Abdominal circumference | Baseline, 5 and 10 months
  Metallic tape measure
Number of participants with adverse events or damages | Baseline, 5 and 10 months
  A self-designed questionnaire consisting of categorical questions (yes or no) will be utilized to assess adverse events. The severity of adverse events will be graded using version 5.0 of the "Common Terminology Criteria for Adverse Events" (CTCAEv5.0). Possible adverse events related to the intervention will be documented in the questionnaire.
Change in baseline Falls Efficacy Scale-International at ten months | Baseline, 5 and 10 months
  The risk of falling will be assessed by means of the Falls Efficacy Scale-International (FES-I) questionnaire in its Brazilian version, which evaluates the concern with the possibility of falling when performing 16 activities, with respective scores from one to four. The total score can vary from 16 (no concern) to 64 (extreme concern).
Change in baseline Berg Balance Scale at ten months | Baseline, 5 and 10 months
  Test: The Berg Balance Scale (BBS) assesses functional balance in the elderly, identifying the risk of falls and monitoring rehabilitation interventions. Composed of 14 items related to daily activities, such as getting up from a chair or turning, the scale uses a score from 0 to 4 for each item, resulting in a maximum total score of 56 points. Interpretive scales include: 0-20 (high risk of falls), 21-40 (moderate risk) and 41-56 (low risk). It is easy to administer, requires little equipment and takes around 15 minutes.
Change in baseline Fatigue Symptom Inventory at ten months | Baseline, 5 and 10 months
  The Fatigue Symptom Inventory (FSI), in its Brazilian version, is a 14-item self-report measure designed to assess the severity, frequency and daily pattern of fatigue, as well as its interference with quality of life. Severity is measured on separate 11-point scales (0=not at all fatigued; 10=as fatigued as possible) that assess the greatest, least and average fatigue in the previous week, as well as current fatigue. Frequency is measured as the number of days in the past week (0-7) on which respondents felt fatigued, as well as the average duration of each day on which they felt fatigued (0=no day; 10=the whole day). Perceived interference is measured on separate 11-point scales (0=no interference; 10=extreme interference) that assess the degree to which fatigue in the previous week interfered with the general level of activity, ability to bathe and dress, normal work activity, ability to concentrate, relationships with others, enjoyment of life and mood.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Costa Moreira, Study Director — Federal University Of Viçosa; Edison A Pérez Bedoya, Study Director — Antioquia University
Locations (2):
- Brazil (2):
  - Universidade Federal de Viçosa, Viçosa, Minas Gerais
  - Federal University of Viçosa, Viçosa - Minas Gerais, Viçosa, Minas Gerais

IPD SHARING:
Plan to Share IPD: No